CLINICAL TRIAL: NCT02399839
Title: Global Lomitapide Pregnancy Exposure Registry
Status: Terminated | Type: Observational
Why Stopped: The PER objective has been integrated into the LOWER protocol.
Sponsor: Amryt Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: AEGR-733-027
Record Dates: First submitted 2015-03-23; First posted 2015-03-26 (Estimated); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Pregnancy
MeSH Terms: interventions — BMS201038

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: lomitapide — As prescribed by Physician.
  Other Names: Juxtapid; Lojuxta

SUMMARY:
To evaluate the outcomes of pregnancy in women treated with lomitapide.

DETAILED DESCRIPTION:
To evaluate the outcomes of pregnancy in women treated with lomitapide at any time within 30 days prior to first day of Last Menstrual Period (LMP) or during pregnancy. The outcomes of primary interest are major congenital anomalies.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant females exposed to lomitapide at any time within 30 days prior to first day of the LMP or during pregnancy.

Exclusion Criteria:

* Patients who are unable or unwilling to provide written informed consent or assent are not eligible to participate in the PER.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant Females
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2014-10; Primary Completion 2022-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Pregnancy | 2 Years
  To evaluate the outcomes of pregnancy in women treated with lomitapide at any time within 30 days prior to first day of Last Menstrual Period (LMP) or during pregnancy. The outcomes of primary interest are major congenital anomalies.

CONTACTS AND LOCATIONS:
Overall Officials: Sallyann O'Brien, Study Director — Amryt Pharmaceuticals
Locations (1):
- Klinikum der Universität München, München, Bavaria, Germany